CLINICAL TRIAL: NCT01921400
Title: The Pathogenesis of Hepatitis C Virus Vertical Transmission
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Maryland (Other); Cairo University (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-0958
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Hepatitis C; Infection Transmission, Maternal-Fetal
Keywords: Hepatitis C (HCV); Infection Transmission, Maternal-Fetal; Placenta; Trophoblast
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Our planned protocol will be to secure whole placental organs after delivery for study patients. Tissue preparation will include a combination of segments preserved in nucleic acid preservative (TriZol or equivalent) and flash freeze of sections to preserve cellular anatomy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HCV-infected mothers: in situ hybridization
- Uninfected mothers: in situ hybridization

SUMMARY:
To evaluate for the presence of HCV Core protein, HCV RNA and SPP in the placenta and fetal membranes using paraffin-embedded sections and post-delivery specimens respectively. In parallel, we will assess placental tissue for evidence of HCV infection using a novel in situ hybridization technique and translate our in vitro findings to these in vivo samples.

Our overall hypothesis is that cytotrophoblasts at the maternal-fetal interface within the placenta serve as a "barrier" that must be crossed during vertical transmission and that cytotrophoblasts are permissive to HCV at a low level that may be enhanced under certain conditions. By comparing the regulation of key steps in the intracellular life cycle of HCV in cytotrophoblasts to highly permissive hepatocytes, significant differences in HCV regulation should be revealed.

Based on our preliminary data, our working hypothesis is that HCV Core protein is differentially processed in cytotrophoblasts compared to hepatocytes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with HCV infection
* Pregnant women without HCV infection

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with HCV infection who present to our collaborating institution in Egypt, and at UNC
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To evaluate for the presence of HCV Core protein, HCV RNA and SPP in the placenta and fetal membranes using paraffin-embedded sections and post-delivery specimens respectively. | 1 year
  We will begin by examining paraffin-embedded sections from HCV-infected mothers who had the placentas sent to pathology for analysis.We will perform a combination of immunohistochemistry (IHC) and immunofluorescence (IF) to analyze the level of SPP expression in the trophoblast cell layer, as well as if HCV Core protein expression was detectable in this layer or in any cell type within the placental section.
  We would also plan to identify other patient-derived tissues that were not paraffin embedded, both from uninfected patients and infected patients to validate different parts of our preliminary data. We would plan to use dissected fetal membranes, which contain both chorion and amnion, to investigate the level of SPP expression in these tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Jhaveri, M.D., Principal Investigator — UNC Department of Pediatrics: Division of Allergy, Immunology, Rheumatology and Infectious Diseases
Locations (2):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States
- Cairo University, Giza, Egypt

REFERENCES:
- [Result] Jhaveri R, Hashem M, El-Kamary SS, Saleh DA, Sharaf SA, El-Mougy F, Abdelsalam L, Ehab M, El-Ghazaly H. Hepatitis C Virus (HCV) Vertical Transmission in 12-Month-Old Infants Born to HCV-Infected Women and Assessment of Maternal Risk Factors. Open Forum Infect Dis. 2015 Jun 26;2(2):ofv089. doi: 10.1093/ofid/ofv089. eCollection 2015 Apr. PMID 26180831